CLINICAL TRIAL: NCT04283019
Title: The Pharmacokinetic and Pharmacodynamic Effects of Oral Cannabidiol (CBD) Under Acute and Chronic Exposure Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Substance Abuse And Mental Health Administration (Unknown); Canopy Growth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00239558
Record Dates: First submitted 2020-02-06; First posted 2020-02-25 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Cannabis, Drug Effects
Keywords: Cannabidiol
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Participants (N=60), will be randomized to 1 of 3 oral dosing conditions that include: 100mg CBD/3.7mg THC (0.39% THC), 100mg CBD/2.8mg THC (0.3% THC), or 100mg CBD/0mg THC (0.0% THC).
Who Masked: Participant, Outcomes Assessor
Masking Description: dosing will be double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CBD without THC (Experimental): oral formulation containing 100mg CBD and 0mg THC
  Interventions: Drug: CBD
- CBD with 3.7 mg THC (Experimental): oral formulation containing 100mg CBD and 3.7mg THC
  Interventions: Drug: CBD; Drug: THC
- CBD with 2.8 mg THC (Experimental): oral formulation containing 100mg CBD and 2.8 mg THC
  Interventions: Drug: CBD; Drug: THC

INTERVENTIONS:
Drug: CBD — CBD will be orally ingested
Drug: THC — THC will be orally ingested
  Arms: CBD with 2.8 mg THC; CBD with 3.7 mg THC

SUMMARY:
This study will evaluate the pharmacokinetic and pharmacodynamic effects of oral Cannabidiol (with or without low levels of THC), under acute and chronic dosing conditions.

DETAILED DESCRIPTION:
Participants (N=60), will be randomized to 1 of 3 oral dosing conditions that include: 100mg CBD/3.7mg THC (0.39% THC), 100mg CBD/2.8mg THC (0.3% THC), or 100mg CBD/0mg THC (0.0% THC). Participants will first complete an 8-hour drug administration session and after this initial session, participants will take participants' assigned study drug for the next 14 days at home, twice daily (participants will visit the lab on days 2, 7, and 14). Participants will return on day 21 (after 1 week washout) for a final visit. During the 8-hour session and visits occurring during the following 21 days, participants will provide biospecimens (urine, blood, oral fluid, hair) which will be tested for cannabinoid concentrations. Pharmacodynamic assessments (subjective and cognitive effects) will also be assessed during these visits.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent
2. Be between the ages of 18 and 55
3. Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests
4. Test negative for recent cannabis use in urine at the screening visit and again upon admission for each experimental session
5. Test negative for other drugs of abuse, including alcohol at the screening visit and upon arrival for each experimental session
6. Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at clinic admission.
7. Have a body mass index (BMI) in the range of 19 to 36 kg/m2
8. Have head hair that is at least 4 cm (approximately one and a half inches) in length on the back of the head.
9. Blood pressure at Screening Visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
10. Report prior experience using cannabis or CBD.
11. Have not donated blood in the prior 30 days.
12. Have a smartphone capable of downloading/operating the Redcap mobile application.

Exclusion Criteria:

1. Non-medical use of psychoactive drugs other than, nicotine, alcohol, or caffeine in the month prior to the screening visit.
2. History of or current evidence of significant medical or psychiatric illness judged by the investigator to put the participant at greater risk of experiencing an adverse event due to exposure or completion of other study procedures.
3. Use of an over-the-counter (OTC), systemic or topical drug(s), herbal supplement(s), or vitamin(s) within 14 days of study entry; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
4. Use of a prescription medication (with the exception of birth control prescriptions) within 14 days of study entry; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject. This includes any medication metabolized via CYP2D6, CYP2C9, CYP2B10, or which induce/inhibit CYP3A4 enzymes.
5. Use of hemp seeds or hemp oil in any form in the past 3 months.
6. Use of dronabinol (Marinol) within the past 6 months.
7. History of xerostomia (dry mouth), or the presence of mucositis, gum infection or bleeding, or other significant oral cavity disease or disorder that in the investigator's opinion may affect the collection of oral fluid samples.
8. History of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina).
9. Enrolled in another clinical trial or have received any drug as part of a research study within 30 days prior to dosing.
10. Epilepsy or a history of seizures.
11. Individuals who have a recent history of traumatic brain injury diagnosed by CT/MRI and have current sequela from prior brain injury, as determined by the study physician
12. Individuals with anemia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Urine cannabinoids | Day 1, 2, 7, 14, and 21
  Concentration of cannabinoids will be measured in urine (unit of measurement: nanograms/mL)

SECONDARY OUTCOMES:
Subjective drug effects as assessed by the Drug Effect Questionnaire | Day 1
  Subjective drug effect ratings (0-100) will be collected with the Drug Effect Questionnaire, with 0 being no effect and 100 being maximum effect.
Subjective drug effects as assessed by the Drug Effect Questionnaire | Day 2
  Subjective drug effect ratings (0-100) will be collected with the Drug Effect Questionnaire, with 0 being no effect and 100 being maximum effect.
Subjective drug effects as assessed by the Drug Effect Questionnaire | Day 7
  Subjective drug effect ratings (0-100) will be collected with the Drug Effect Questionnaire, with 0 being no effect and 100 being maximum effect.
Subjective drug effects as assessed by the Drug Effect Questionnaire | Day 14
  Subjective drug effect ratings (0-100) will be collected with the Drug Effect Questionnaire, with 0 being no effect and 100 being maximum effect.
Subjective drug effects as assessed by the Drug Effect Questionnaire | Day 21
  Subjective drug effect ratings (0-100) will be collected with the Drug Effect Questionnaire, with 0 being no effect and 100 being maximum effect.
Blood cannabinoids | Day 1, 2, 7, 14, and 21
  Concentration of cannabinoids will be measured in blood (unit of measurement: nanograms/mL)
Oral Fluid cannabinoids | Day 1, 2, 7, 14, and 21
  Concentration of cannabinoids will be measured in oral fluid (unit of measurement: nanograms/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No